CLINICAL TRIAL: NCT03626454
Title: Efficacy and Safety of Prophylactic Norepinephrine Addition in Prevention of Hypotension During Spinal Anesthesia for Caesarean Delivery: A Randomized Trial
Brief Title: Norepinephrine Addition in Spinal Anesthesia of Caesarean Section
Acronym: NASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Yasser S Mostafa, MD, Lecturer of anesthesia, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NASA2018
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hypotension Drug-Induced
Keywords: Norepinephrine, hypotension, spinal, caesarean section
MeSH Terms: conditions — Hypotension | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: An anesthesia resident who will not be involved with the conduct of the study will prepare and label the drug in the syringes according to the randomization codes.
  An investigator who will not be involved in subsequent patient care or assessment will open the topmost of 300 opaque sequentially numbered envelopes. One 50 ml and one 10 ml will be labeled as study drug and the 50 ml syringe will be connected to a syringe infusion pump. These two "study drug" syringes will be a part of double dummy technique to facilitate blindness. In group B, 50 ml syringe will contain saline, and 10 ml syringe will contain norepinephrine (.6 µg/ml). In group I, 50 ml syringe will contain norepinephrine (6 µg/ml) with, and 10 ml syringe will contain saline. Participant in both groups will receive bolus from 10 ml syringe over 30 seconds and infusion dose of 1 ml/kg/h simultaneously to expedite blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group B (Active Comparator): 'Norepinephrine bolus' of 6 µg plus Normal Saline 0.9% Infusion Solution
  Interventions: Drug: Norepinephrine Bolus; Drug: Normal Saline 0.9% Infusion Solution
- group I (Active Comparator): 'Norepinephrine infusion' 6 µg/kg/h plus 'Normal Saline Flush, 0.9% Injectable Solution
  Interventions: Drug: Norepinephrine infusion; Drug: Normal Saline Flush, 0.9% Injectable Solution

INTERVENTIONS:
Drug: Norepinephrine Bolus — 'Norepinephrine Bitartarte' bolus of 6 µg/mL for 30 seconds immediately after intrathecal injection
  Other Names: NORB
  Arms: group B
Drug: Norepinephrine infusion — an infusion of 6 µg/mL norepinephrine that was started at 6 µg/kg/h immediately after intrathecal injection
  Other Names: NORI
  Arms: group I
Drug: Normal Saline Flush, 0.9% Injectable Solution — 10 ml normal saline in syringe for bolus for 30 seconds immediately after intrathecal injection
  Other Names: NORSB
  Arms: group I
Drug: Normal Saline 0.9% Infusion Solution — 50 ml syringe with normal saline infuse at a rate 1ml/kg/h immediately after intrathecal injection
  Other Names: NORSI
  Arms: group B

SUMMARY:
The objective is to compare efficacy of prophylactic norepinephrine bolus versus Infusion in prevention of hypotension which occurs frequently after spinal anesthesia for caesarean section. The authors hypothesize that prophylactic norepinephrine bolus is as effective as infusion in Prevention of hypotension after spinal anesthesia in caesarean section

DETAILED DESCRIPTION:
Introduction Spinal anesthesia is the technique of choice for elective cesarean delivery. During spinal anesthesia for cesarean delivery, maternal hypotension is a major complication with the incidence up to 60-70%. Prolonged hypotension leads to decreased utero-placental blood flow and fetal acidosis. Vasopressors such as ephedrine, phenylephrine, and norepinephrine are therefore commonly recommended to reduce the incidence of hypotension.Phenylephrine is currently the first-choice vasopressor for prevention and treatment of maternal hypotension during spinal anesthesia for cesarean delivery (CD).

phenylephrine in this context has been questioned, owing to its propensity to increase afterload, reduce maternal heart rate, and reduce cardiac output. A recent studies indicated that norepinephrine infusion or bolus during spinal anesthesia for cesarean delivery was associated with greater heart rate and cardiac output compared with phenylephrine. Other studies also showed that norepinephrine could act as an alternative to phenylephrine without adverse outcomes.Because it is a potent α-adrenergic agonist with some β-adrenergic effect and, therefore, should not have a tendency to reduce heart rate and cardiac output as much as phenylephrine.

The use of norepinephrine to prevent and treat hypotension during CD is new and data in the literature are scarce. Although treatment of hypotension during spinal anesthesia is listed by the manufacturer as an indication for the use of norepinephrine, there is limited information available for its use for this purpose in the literature and few reports of its use in obstetric patients.

Carvalho and Dyer suggested that more investigations of norepinephrine using simpler methods of delivery than computer-controlled systems are required. Such studies are now emerging.

Anesthetic technique:

Patients will fast overnight and no premedication will be administered. On the day of surgery in the operating room, intravenous (IV) access will be obtained with an 18 gauge IV cannula in an upper limb vein and an infusion of lactated Ringer's (LR) solution of 10 ml/kg will be started as a bolus immediately preceding and with the intrathecal injection, followed by a maintenance rate of 15-30 ml/minute to keep the vein open until delivery of the fetus. Infusion bags will be suspended approximately 1.5 meter above the mid-point of the top surface of the operating table, and the fluid will be administered through a wide-bore administration set with the clamp fully opened.

All patients will be monitored by standard routine monitoring which includes a 5-lead electrocardiography, a non-invasive blood pressure, pulse oximetry. A baseline systolic blood pressure (SBP), mean arterial pressure (MAP) and heart rate (HR) will be measured and recorded in the sitting position by averaging 3 readings taken 1 minute apart using an automated device for noninvasive blood pressure assessment and pulse oximetry (or electrocardiography). All measurements will be continuously recorded until the end of surgery and to avoid possible influence on the measurements, the monitoring module will be placed on the other arm of IV cannula. Spinal anesthesia will be performed with the patient in the sitting position, using a 25-gauge Quincke needle after full aseptic precautions. After skin infiltration with lidocaine 2% (w/v), spinal needle will be inserted at what will be estimated to be the L3 to L4 or L4 to L5 vertebral interspace. After confirmation of free flow of cerebrospinal fluid, intrathecal injection using 0.5% hyperbaric bupivacaine 2.2-2.5 ml mixed with preservative-free fentanyl 15 µg will be injected over 15 seconds, as per our standard practice to achieve surgical anesthesia. The patient will be then positioned supine, with left uterine displacement using a wedge under the right hip. Oxygen 3 L/min via nasal prongs or 5 L/min via mask, if the oxygen saturation fell below 95%. Block level will be assessed by pinprick with a 23 G needle and controlled within T4-6.

Immediately after intrathecal injection, the study medications will be started at 1 ml/kg/h using an infusion pump and injected for 30 seconds for bolus. A rescue bolus of 10 µg norepinephrine or 15 mg ephedrine will be used to treat hypotension. The study protocol will be continued until the end of surgery. After delivery, intravenous oxytocin of 15 U will be administered by slow infusion.

The time interval between blood pressure readings will be 1 minute, therefore the maximum frequency of administration of norepinephrine will be every minute. Hypotension will be defined as a SBP < 80% of the baseline value, in which case the treatment will be deemed a failure, and the anesthesiologist in charge will revert to the standard practice ephedrine 5 mg/mL. Hypertension will be defined as a SBP > 120% of the baseline value, in which case the study solution will be held until the SBP will be less than baseline and a vasodilator (nitroglycerin) can be given if necessary. Bradycardia will be defined as a heart rate < 50 bpm and can be treated with anticholinergics (0.6 mg atropine) if necessary. Decision to treat will be at the discretion of the anesthesiologist. All patients with sensory block levels lower than T6 at 20 minutes were to be considered a dropout.

Use of norepinephrine after completion of the study period will be at the discretion of the attending anesthesiologist, otherwise ephedrine 5 mg/mL will be used, as per standard practice. Upon delivery, a segment of the umbilical cord will be collected for assessment of blood gases in both the umbilical artery and umbilical vein. Hemodynamic values including SBP, MBP, DBP and HR will be recorded at the following timepoints: baseline, after 3 minutes, 5 minutes, 10 minutes, 15 minutes, 20 minutes (± 30 minutes), delivery of fetus, oxytocin administration and end of surgery. Norepinephrine consumption before delivery and during the surgery will be recorded. Adverse effects including shivering, headache, restlessness, pruritus, and peripheral vascular constriction will be recorded. In addition, neonatal outcomes including umbilical venous blood gases and Apgar scores at 1 and 5 min will be recorded by the attending pediatrician, who will be unaware of the vasopressor used

Statistical analysis:

For Sample size calculation MedCalc Statistical Software version 18 (MedCalc Software bvba, Ostend, Belgium; http://www.medcalc.org; 2018) is used. According to previous studies showing that incidence of hypotension among norepinephrine bolus 15% is while it is 31% among norepinephrine infusion. So, a sample size of 144 patients per group will be required to detect a difference of 16% with allocation ratio 1, two-sided α error of 0.05 and 90% power. To compensate for possible dropouts or excluded cases, the authors will include 150 patients in each group with total sample size of 300 patients. Statistical analysis will be performed using SPSS version 24.0 (IBM, Armonk, NY, USA). Data will be tested for normality using the Kolmogorov-Smirnov test. Continuous variables are presented as mean ± standard deviation (SD) or median (interquartile range) as appropriate and categorical variables are presented as number of patients (%). Parametric continuous variables will be analyzed by unpaired t-test and non-parametric continuous variables will be analyzed by Mann-Whitney U test. For categorical variables, the Chi-square (X2) test or Fisher's exact test will be used as appropriate. Two-tailed p values of 0.05 will be considered statistically significant.For Sample size calculation MedCalc Statistical Software version 18 (MedCalc Software bvba, Ostend, Belgium; http://www.medcalc.org; 2018) is used. Previous studies show that the incidence of hypotension among norepinephrine bolus 15% is while it is 31% among norepinephrine infusions. So, a sample size of 105 patients per group will be required to detect a difference of 16% with allocation ratio 1, two-sided α error of 0.05, and 80% power. To compensate for possible dropouts or excluded cases, the authors will include 110 patients in each group with a total sample size of 220 patients. Statistical analysis will be performed using SPSS version 24.0 (IBM, Armonk, NY, USA). Data will be tested for normality using the Kolmogorov-Smirnov test. Continuous variables are presented as mean ± standard deviation (SD) or median (interquartile range) as appropriate and categorical variables are presented as number of patients (%). Parametric continuous variables will be analyzed by unpaired t-test and non-parametric continuous variables by Mann-Whitney U test. The Chi-square (X2) test or Fisher's exact test will be used as appropriate for categorical variables. Two-tailed p-values of 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years
* American Society of Anesthesiologists physical status classification II or III
* Elective caesarean section under spinal anesthesia
* Normal singleton pregnancy beyond 36 weeks gestation
* Weight 50-100 kg, height 150-180 cm

Exclusion Criteria:

* Patient refusal
* Allergy or hypersensitivity to norepinephrine
* Diabetes, excluding gestational diabetes
* Preexisting or pregnancy-induced hypertension
* Arrhythmia
* Cerebrovascular disease
* Known fetal abnormality or fetal distress
* Any contraindication to spinal anesthesia
* Use of monoamine oxidase inhibitors, triptyline or imipramine antidepressants

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | 5 to 15 minutes after giving spinal anesthesia
  less than 80% baseline blood pressure

SECONDARY OUTCOMES:
Baseline heart rate | 3 minutes before giving spinal anesthesia
  in beats/min
Baseline mean blood pressure | 3 minutes before giving spinal anesthesia
  in mmHg
Baseline systolic blood pressure | 3 minutes before giving spinal anesthesia
  in mmHg
Anesthesia to delivery time | from immediately after giving anesthesia until delivery of fetus by surgeon
  in minutes
Incision to delivery time | in time of beginning of surgical incision of skin until delivery of fetus by surgeon
  in minutes
Uterine incision to delivery time | in time of beginning of uterine incision until delivery of fetus by surgeon
  in seconds
Presence of Nausea | 30 minutes
  Presence of nausea in patients from induction of spinal anesthesia to delivery of the fetus.
Presence of vomiting | 30 minutes
  Presence of vomiting in patients from induction of spinal anesthesia to delivery of the fetus.
Incidence of hypertension | 30 minutes
  Systolic blood pressure at or above 120% of baseline, from induction of spinal anesthesia to delivery of the fetus
Occurence of bradycardia | 30 minutes
  Heart rate less than 50 bpm, from induction of spinal anesthesia from induction of spinal anesthesia to delivery of the fetus
Occurence of tachycardia | 30 minutes
  Heart rate more than 120 bpm, from induction of spinal anesthesia from induction of spinal anesthesia to delivery of the fetus
Upper sensory level of anesthetic block | 3 minutes after giving spinal anesthesia
  assessment by pin prick
Umbilical artery pH | 1 minute after delivery
  from umbilical artery blood gases
Umbilical vein pH | 1 minute after delivery
  from umbilical vein blood gases
Umbilical artery partial pressure of carbon dioxide | 1 minute after delivery
  from umbilical artery blood gases
Umbilical vein partial pressure of carbon dioxide | 1 minute after delivery
  from umbilical vein blood gases
Umbilical artery partial pressure of oxygen | 1 minute after delivery
  from umbilical artery blood gases
Umbilical vein partial pressure of oxygen | 1 minute after delivery
  from umbilical vein blood gases
Umbilical artery bicarbonate | 1 minute after delivery
  from umbilical artery blood gases
Umbilical artery base excess | 1 minute after delivery
  from umbilical artery blood gases
Umbilical vein bicarbonate | 1 minute after delivery
  from umbilical vein blood gases
Umbilical vein base excess | 1 minute after delivery
  from umbilical vein blood gases
APGAR score | 1 minute after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 minutes after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
Rescue ephedrine dose | every 2 minutes up to 30 minutes immediately after occurence of hypotension
  10 mg given intravenous
first rescue ephedrine dose time | 1 minute after giving rescue ephedrine
  in min
Total used ephedrine dose | 1 minute after correction of blood pressure
  in mg

OTHER OUTCOMES:
Age | 1 hour before operation once the patient recruited
  in years
Weight | 1 hour before operation once the patient recruited
  In kilograms
Height | 1 hour before operation once the patient recruited
  In meters
BMI | 1 hour before operation once the patient recruited
  In kilogram per square meter
Gestational age | 1 hour before operation once the patient recruited
  in weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hany M Yassin, M.D., Study Chair — Fayoum University
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Khaw KS. Prophylactic Norepinephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery. Anesth Analg. 2018 Jun;126(6):1989-1994. doi: 10.1213/ANE.0000000000002243. PMID 28678073
- [Background] Onwochei DN, Ngan Kee WD, Fung L, Downey K, Ye XY, Carvalho JCA. Norepinephrine Intermittent Intravenous Boluses to Prevent Hypotension During Spinal Anesthesia for Cesarean Delivery: A Sequential Allocation Dose-Finding Study. Anesth Analg. 2017 Jul;125(1):212-218. doi: 10.1213/ANE.0000000000001846. PMID 28248702
- [Background] Ngan Kee WD, Khaw KS, Tan PE, Ng FF, Karmakar MK. Placental transfer and fetal metabolic effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology. 2009 Sep;111(3):506-12. doi: 10.1097/ALN.0b013e3181b160a3. PMID 19672175
- [Background] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Background] Chen D, Qi X, Huang X, Xu Y, Qiu F, Yan Y, Li Y. Efficacy and Safety of Different Norepinephrine Regimens for Prevention of Spinal Hypotension in Cesarean Section: A Randomized Trial. Biomed Res Int. 2018 May 23;2018:2708175. doi: 10.1155/2018/2708175. eCollection 2018. PMID 29951531
- [Background] Carvalho B, Dyer RA. Norepinephrine for Spinal Hypotension during Cesarean Delivery: Another Paradigm Shift? Anesthesiology. 2015 Apr;122(4):728-30. doi: 10.1097/ALN.0000000000000602. No abstract available. PMID 25654435